CLINICAL TRIAL: NCT07275710
Title: Role of Alprazolam in Management of Post Endodontic Pain After Single Visit Root Canal Treatment
Brief Title: Role of Alprazolam in Management of Post Endodontic Pain After Single Visit Root Canal Treatment. To Compare Mean Pain Score Between Two Group of Participants Undergoing Post Operative Pain Management After Single Visit Root Canal Treatment: NSAIDs Alone and a Combination of NSAIDs and Alprazolam.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Armed Forces Post Graduate Medical Institute (AFPGMI), Rawalpindi (Other)
Responsible Party: Principal Investigator, Tahreem Qureshi, Principal Investigator, Armed Forces Post Graduate Medical Institute (AFPGMI), Rawalpindi
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: OD2025-PAIN-01
Record Dates: First submitted 2025-11-16; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Pain
Keywords: post endodontic pain; root canal treatment; alprazolam
MeSH Terms: conditions — Pain | interventions — Ibuprofen; Alprazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- brufen (Active Comparator): one group in the study will be prescribed 400mg ibuprofen tablet for management of post endodontic pain after root canal treatment and patient will be asked to score their pain level at 6, 12 and 24 hours on visual analogue scale.
  Interventions: Drug: Brufen
- alprazolam (Active Comparator): second group in the study will be prescribed 0.5mg alp tablet for management of post endodontic pain after root canal treatment and patient will be asked to score their pain level at 6, 12 and 24 hours on visual analogue scale.
  Interventions: Combination Product: Brufen and alprazolam

INTERVENTIONS:
Combination Product: Brufen and alprazolam — second group in the study will be prescribed 400mg ibuprofen and 0.5mg alp tablet for management of post endodontic pain after root canal treatment
  Arms: alprazolam
Drug: Brufen — one group in the study will be prescribed 400mg ibuprofen for management of post endodontic pain after root canal treatment
  Arms: brufen

SUMMARY:
To compare mean pain score between two group of participants undergoing post operative pain management after single visit root canal treatment: one group receiving NSAIDs alone and the other receiving a combination of NSAIDs and an anxiolytic medication i.e alprazolam.

DETAILED DESCRIPTION:
This randomized controlled clinical trial is designed to compare postoperative pain levels following single-visit root canal treatment in patients receiving two different analgesic regimens: ibuprofen alone or a combination of ibuprofen and alprazolam.

Eligible patients will be screened through detailed medical and dental histories, clinical examinations, and necessary diagnostic tests, including periapical radiographs. Participants meeting the inclusion criteria will be divided into two equal groups using a scientific random number table to ensure unbiased allocation. Matching will be performed based on relevant variables such as age, gender, and tooth location to minimize confounding factors.

Root canal therapy will be carried out in a single visit under local anesthesia (Septodent, Lignospan Special; 2% lignocaine hydrochloride with 1:80,000 adrenaline) and rubber dam isolation. The working length will be determined 1 mm short of the radiographic apex using an apex locator (DENTSPLY Maillefer, Denta Port ZX) and verified radiographically.

Canal instrumentation will be performed with ProTaper Universal hand files (DENTSPLY Sirona) under copious irrigation with 5.25% sodium hypochlorite solution (Henry Schein). Instrumentation will proceed up to F2 ProTaper size. Canal patency will be maintained using a #10 K-file (DENTSPLY Maillefer) between each instrument change. A final rinse with 17% EDTA (ERKAMED Endo-Prep Gel) will be used to remove the smear layer.

After chemo-mechanical preparation, canals will be dried with sterile paper points (Sure-Endo). Obturation will be performed using the single-cone technique with F2 gutta-percha points (Bio GP Points, Sure-Endo) and endodontic sealer (President Dental Germany, Endoplus). The master cone position will be confirmed radiographically. Sealer placement will be accomplished with a lentulospiral (DENTSPLY Sirona) in a slow-speed handpiece. All clinical procedures will be completed by a single operator in one visit. After obturation, the access cavity will be sealed with a 4 mm thickness of temporary filling material (DETAX, Fermin). Patients will be recalled after one week for permanent restoration.

Blinding

To minimize bias, blinding will be implemented at multiple levels:

* Patient Blinding: Patients will be unaware of the specific drug comparison and will be informed only that the study evaluates postoperative pain following root canal therapy.
* Operator Blinding: A single operator will perform all treatments but will not participate in postoperative pain assessment.
* Outcome Assessor Blinding: The evaluator responsible for collecting pain scores and performing statistical analysis will be blinded to group assignments.

Intervention Groups

Following completion of obturation and placement of the temporary restoration, patients will be randomly assigned to one of two groups:

* Group 1: Ibuprofen 400 mg (Abbott Brufen)
* Group 2: Ibuprofen 400 mg (Abbott Brufen) + Alprazolam 0.5 mg (Hilton Pharma Alp)

Pain Assessment

Participants will be provided with a pain diary containing a 10 cm Visual Analogue Scale (VAS) ranging from 0 (no pain) to 10 (worst possible pain). They will record their pain intensity at 6, 12, and 24 hours after treatment. Pain diaries will be collected during the one-week follow-up visit. Data will be used to compare mean VAS scores between groups to evaluate the efficacy of the two analgesic regimens.

ELIGIBILITY:
Inclusion Criteria:

* patients aged between 18-60 years
* healthy patients with ASA classification I and II
* Teeth with symptomatic irreversible pulpitis

Exclusion Criteria:

* patient suffering from systemic disease that requires antibiotics
* pregnant or lactating mothers
* teeth with periapical radiolucency
* teeth with severe periodontitis
* patients who have taken analgesics 12 hours prior to procedure
* patients already taking benzodiadepines

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
pain levels | 6 hours 12 hours 24 hours
  patients will be randomly assigned to one of two groups:
  * Group 1: Ibuprofen 400 mg (Abbott Brufen)
  * Group 2: Ibuprofen 400 mg (Abbott Brufen) + Alprazolam 0.5 mg (Hilton Pharma Alp)
  Pain Assessment
  Participants will be provided with a pain diary containing a 10 cm Visual Analogue Scale (VAS) ranging from 0 (no pain) to 10 (worst possible pain). They will record their pain intensity at 6, 12, and 24 hours after treatment. Pain diaries will be collected during the one-week follow-up visit. Data will be used to compare mean VAS scores between groups to evaluate the efficacy of the two analgesic regimens.

CONTACTS AND LOCATIONS:
Locations (1):
- Armed Forces Post Graduate Medical Institute, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study does not include plans or infrastructure for secure long-term data storage, de-identification, and controlled access needed to protect participant privacy. Additionally, the dataset is small, and disclosure may increase the risk of re-identification. Summary results will be made available as required.

REFERENCES:
- [Background] Baradaran M, Hamidi MR, Moghimi Firoozabad MR, Kazemi S, Ashrafpour M, Moghadamnia AA. Alprazolam role in the analgesic effect of ibuprofen on postendodontic pain. Caspian J Intern Med. 2014 Fall;5(4):196-201. PMID 25489429

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-11-15): https://cdn.clinicaltrials.gov/large-docs/10/NCT07275710/Prot_SAP_ICF_000.pdf